CLINICAL TRIAL: NCT02599233
Title: Characterization of Post-operative Pain Trajectories Over Seven Days and Their Potential Links With Chronicity After 3 Months: a Single-center, Prospective, Pilot Cohort Study at the Nîmes University Hospital
Brief Title: Characterization of Post-operative Pain Trajectories Over Seven Days and Links With Chronicity
Acronym: PATCH
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2015/JLH-01; 2015-A00868-41 (Other: ANSM)
Record Dates: First submitted 2015-11-04; First posted 2015-11-06 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2017-01

CONDITIONS: Surgical Procedures, Operative; Pain; Chronic Pain
Keywords: pain trajectory
MeSH Terms: conditions — Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- The study population: The study population consists of adult surgery patients at the Nîmes University Hospital, with recruitment based on the operating theater program for a predefined six month period and for a predefined list of surgeries. The latter list of surgical acts was established according to the Medicalization of Information Systems Progam (PMSI) database. Patients are recruited either the day before or the day after surgery, in their respective departments.
  Interventions:
  * In hospital pain evaluation
  * In hospital questionnaires
  * Telephone conctact at 3 months
  Interventions: Other: Telephone conctact at 3 months; Other: In hospital pain evaluation; Other: In hospital questionnaires

INTERVENTIONS:
Other: Telephone conctact at 3 months — Patients will be contacted at 3 months post-surgery for pain questionnaires.
Other: In hospital pain evaluation — Patients will evaluate their pain levels via a verbal numerical scale on days 1(or-1), 2, 3, 4, 5, 6 & 7.
Other: In hospital questionnaires — Patients are required to fill out the HADS and PCS questionnaires between on day -1 or +1.

SUMMARY:
The main objective of this study is to establish the postoperative "pain pathways" observed from D1 to D7 in the context of the current management after orthopedic, digestive, obstetrics and gynecology, urology, neurosurgery, vascular and thoracicn surgeries.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A. To assess the incidence of Post-Surgical Chronic Pain (PSCP) Chronic 3 months post intervention.

B. To asses the incidence of neuropathic type pain (DN4 Questionnaire) at 3 months post intervention.

C. To study the potential links between pain trajectories and the presence or absence of PSCP.

D. To study the potential links between the presence or absence of PSCP and known risk factors for PSCP (patient-related data, data on the surgery, anesthesia data).

ELIGIBILITY:
Inclusion Criteria:

* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 3 months of follow-up
* The patient has undergone a planned surgical procedure in one of the participating departments
* The patient is willing and able to respond to the study questionnaires (HADS, PCS, EN, DN4)

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* It is impossible to correctly inform the patient
* Patient admitted to the ICU and still intubated at day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult surgery patients at the Nîmes University Hospital, with recruitment based on the operating theater program for a predefined six month period and for a predefined list of surgeries. The latter list of surgical acts was established according to the Medicalization of Information Systems Progam (PMSI) database. Patients are recruited either the day before or the day after surgery, in their respective departments.
Sampling Method: Probability Sample
Enrollment: 392 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-11-03 (Actual); Study Completion 2016-11-03 (Actual)

PRIMARY OUTCOMES:
The pain trajectory for the first 7 post-operative days. | Day 7 post-surgery
  The pain trajectory is the vector of 7 verbal numerical pain estimates (from 0 to 10) taken over 7 days (days 1 (or -1), 2, 3, 4, 5, 6 & 7).
  Day 0 is the day of surgery.

SECONDARY OUTCOMES:
The DN4 questionnaire | month 3
Since the surgery, do you have persistent pain? yes/no | month 3
Is it the same pain before the surgery? yes/no | month 3
Verbal numberical scale for pain (ranging from 0 to 10) | month 3
Have you had complications from your surgery? yes/no | month 3
Hospital Anxiety and Depression Scale (HADS) | day -1 or day +1
Pain Catastrophizing Scale (PCS) | day -1 or day +1
Cumulative consumption of antalgic drugs | day -1 or day +1
Cumulative consumption of antalgic drugs | day 2
Cumulative consumption of antalgic drugs | day 3
Cumulative consumption of antalgic drugs | day 4
Cumulative consumption of antalgic drugs | day 5
Cumulative consumption of antalgic drugs | day 6
Cumulative consumption of antalgic drugs | day 7

CONTACTS AND LOCATIONS:
Overall Officials: Joël L'Hermite, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

REFERENCES:
- [Result] L'Hermite J, Page MG, Chevallier T, Occean B, Viel E, Bredeau O, Lefrant JY, Cuvillon P. Characterisation of pragmatic postoperative PAin Trajectories over seven days and their association with CHronicity after 3 months: a prospective, pilot cohort study (PATCH study). Anaesth Crit Care Pain Med. 2021 Feb;40(1):100793. doi: 10.1016/j.accpm.2020.100793. Epub 2020 Dec 23. PMID 33359373